CLINICAL TRIAL: NCT02938624
Title: Anti PD-1 Neo-adjuvant Treatment for Early Stage NSCLC - Phase I Study
Brief Title: Anti PD-1 Neo-adjuvant Treatment for NSCLC
Acronym: MK3475-223
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jair Bar, M.D., Ph.D. (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Jair Bar, M.D., Ph.D., Deputy Director, Institute of Oncology, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3282/16SMC
Record Dates: First submitted 2016-10-12; First posted 2016-10-19 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Non Small Cell Lung Carcinoma; Stage I; Stage II
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- cohort1 (Experimental): Pembrolizumab 200 mg I.V single dose
  Interventions: Drug: Pembrolizumab 200 mg IV single dose; Procedure: Surgical resection of tumor
- Cohort II (Experimental): Pembrolizumab 200 mg I.V Twice interval 21 days
  Interventions: Drug: Pembrolizumab 200 mg IV twice interval 21 days; Procedure: Surgical resection of tumor
- Cohort III (Experimental): Pembrolizumab 200 mg IV Twice interval 21d,surgery after 10d
  Interventions: Drug: Pembrolizumab 200 mg IV Twice interval 21d,surgery after 10d; Procedure: Surgical resection of tumor
- COHORT -1 (Experimental): Pembrolizumab 100 mg I.V single dose
  Interventions: Drug: Pembrolizumab 100 mg I.V single dose; Procedure: Surgical resection of tumor

INTERVENTIONS:
Drug: Pembrolizumab 200 mg IV single dose — Pembrolizumab 200 mg IV single dose, 21 days later surgery
  Other Names: keytruda
  Arms: cohort1
Drug: Pembrolizumab 200 mg IV twice interval 21 days — Pembrolizumab 200 mg IV twice interval 21 days, 21 days later surgery
  Other Names: keytruda
  Arms: Cohort II
Drug: Pembrolizumab 200 mg IV Twice interval 21d,surgery after 10d — Pembrolizumab 200 mg IV Twice interval 21d,surgery after 10d
  Other Names: keytruda
  Arms: Cohort III
Drug: Pembrolizumab 100 mg I.V single dose — Pembrolizumab 100 mg I.V single dose, surgery after 21 days.
  Other Names: keytruda
  Arms: COHORT -1
Procedure: Surgical resection of tumor — Surgical resection of tumor by any of the acceptable procedures
  Other Names: Lobectomy/pneumonectomy/bi-lobectomy

SUMMARY:
A single arm, phase I, dose escalation trial and expansion cohort, examining the safety and feasibility of neoadjuvant pembrolizumab treatment for early resectable NSCLC patients.

Hypothesis: The investigators hypothesize that response rate to neo-adjuvant pembrolizumab will be higher than the response rate of advanced NSCLC patients.

DETAILED DESCRIPTION:
16-28 patients with apparently operable NSCLC, clinically staged I-II with a resectable tumor would be recruited. Recruitment would be based on clinical assessment by a qualified Thoracic surgeon, with the appreciation that some of the recruited patients would eventually be deemed to be non-operable, or with a non-resectable disease, or to harbor a diagnosis different from NSCLC.

Screen of consenting patients would include a diagnostic biopsy that includes core needle biopsy procedure. Fresh as well as formalin fixed paraffin embedded baseline tumor samples will be obtained according to common Standard Operating Procedures. Specimens would be processed as per pathology standard of care and two cores or more will be utilized later for the research study.

A patient recruited after a previous diagnostic biopsy, would be eligible for the trial only if willing to undergo a repeat diagnostic procedure as above. Processing of biopsy material will be similar regardless if it is first or second biopsy.

Trial treatment will commence only following pathological confirmation of NSCLC, complete staging including CT-PET and brain imaging, and positive pre-op cardiac and pulmonary assessment.

Study schedule Dose levels of this study are defined by dose of drug as well as number of treatments and required interval from last treatment to surgery. At least 3 subjects in a dose cohort must complete the dose limiting toxicity (DLT) evaluation period before dosing is initiated at the next higher dose level. Only toxicities occurring during the DLT period will be considered as DLTs and utilized to inform dose escalation decisions. The DLT period starts with the first dose of pembrolizumab till 30 days post-surgery.

Cohorts consists of 3-6 subjects per dose level, to be treated with study therapy following a 3+3 schema.

Dose escalation will proceed between cohorts according to a modified "3+3 design," as explained in the following scheme. Dose-limiting toxicity (DLT) is defined below and is confined in time as defined above. As a safety feature, a new dosing/schedule level will open only after the end of 30 post-operative days of the last patient in the previous cohort. If cohort one will be found to be too high as RP2D/schedule, the next patients will be treated at a dose/schedule level minus one. Only one step of dose reduction is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical or pathological diagnosis of early resectable NSCLC stage I-II (AJCC version 7).
2. Have measurable tumor of a least one cm in its largest diameter.
3. Clinically assessed to be a candidate for curative intent lobectomy or larger procedure (e.g. bilobectomy, pneumonectomy, lobectomy with segmentectomy, etc).
4. Is willing to undergo a procedure aimed to collect tumor tissue for pathologic diagnosis and for research correlative studies.
5. Be willing and able to provide written informed consent/assent for the trial.
6. Be > 18 years of age on day of signing informed consent.
7. Have a performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

   Table 1: Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC) >=1,500 /mcL Platelets>=100,000 / mcL Hemoglobin>= 9 g/dL or >=5.6 mmol/L RenalSerum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) <=1.5 X upper limit of normal (ULN) OR >=60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin <=1.5 X ULN OR Direct bilirubin <= ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) <= 2.5 X ULN OR Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants <=1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Severe lung emphysema with a significantly elevated risk of dangerous complications from a biopsy of a lung lesion.
2. Predicted post-operative (PPO)-FEV1 or PPO-DLCO < 30% (as calculated based on patient's age, sex, weight, height and planned operation).
3. Has a known diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., <= Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy (besides as part of a curative treatment for a different malignancy, completed 5 years or more prior recruitment to study).
6. Has a known additional active malignancy. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, low grade bladder TCC or in situ cervical cancer that has undergone potentially curative therapy. History of other malignancies can be permitted provided at least five years have passed since the completion of a potentially curative therapy.
7. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-01-07 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | 24 months
  Protocol defined dose limiting toxicities, aiming to identify RP2D=Recommended Phase 2 Dose/schedule.
Percentage of residual viable tumor cells | 24 months
  Percent residual viable tumor cells in post-treatment pathologic specimen
Percent change in tumor volume | 24 months
  Volumetric CT assessment at CT scan performed prior to surgical resection of tumor, relative to base line CT scan.

SECONDARY OUTCOMES:
Median time-to-recurrence. | 48 Months
  Median time-to-recurrence of disease in NSCLC patients treated with neo-adjuvant pembrolizmab and surgical resection of tumor, assessed by Kaplan-Meier method.
Median Overall survival. | 60 months
  Median Overall survival of NSCLC patients treated with neo-adjuvant pembrolizmab and surgical resection of tumor, assessed by Kaplan-Meier method.

OTHER OUTCOMES:
Change in percentage of cells expressing PDL1 in tumors with treatment | 24 Months
  Comparing pre and post pembrolizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Sheba Medical Centre Jair, MD PHD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No